CLINICAL TRIAL: NCT06203132
Title: Phase III, Open-label, Randomized, Multicenter Trial EvaLuating the Non-inferiority of DORAvirine Versus DOlutegravir Based Antiretroviral Regimens in Treatment-naïve People Living With HIV-1 Infection
Brief Title: DORAvirine Versus DOlutegravir Based Antiretroviral Regimens in Treatment-naïve People Living With HIV-1 Infection
Acronym: ELDORADO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: MSD France (Industry); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 0392s ELDORADO
Record Dates: First submitted 2023-12-06; First posted 2024-01-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: HIV-1-infection
Keywords: HIV-1; ART-naïve; doravirine; dolutegravir; non-inferiority
MeSH Terms: interventions — doravirine; Tenofovir; Lamivudine; dolutegravir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doravirine arm (Experimental): Doravirine (100 mg) + tenofovir DF (300 mg) + lamivudine (300mg) administered daily
  Interventions: Drug: Doravirine + tenofovir DF + lamivudine
- Dolutegravir arm (Active Comparator): Dolutegravir (50 mg) + tenofovir DF 300 mg + XTC (300 mg if lamivudine or 200 mg if emtricitabine) administered daily
  Interventions: Drug: Dolutegravir + tenofovir DF + lamivudine or emtricitabine

INTERVENTIONS:
Drug: Doravirine + tenofovir DF + lamivudine — Oral administration
  Other Names: Delstrigo
  Arms: Doravirine arm
Drug: Dolutegravir + tenofovir DF + lamivudine or emtricitabine — Oral administration
  Arms: Dolutegravir arm

SUMMARY:
Phase III trial evaluating doravirine as an alternative to dolutegravir in treatment naïve people living with HIV-1 infection.

DETAILED DESCRIPTION:
Phase III, multicenter, open-label, randomized, non-inferiority clinical trial which aims to assess the non-inferiority of doravirine in association with tenofovir and lamivudine, as compared to dolutegravir in association with tenofovir and lamivudine or emtricitabine.

This trial will be implemented in Brazil, Cameroon, Côte d'Ivoire, France, Mozambique and Thailand.

Six hundred and ten patients will be enrolled and followed for 96 weeks after entry in the trial (=ART initiation).

Primary endpoint will assess virological efficacy at Week 48, measured by the proportion of subjects achieving HIV-1 RNA <50 copies/mL, in HIV-1 infected, treatment-naive subjects with pre-treatment viral load (HIV-1 RNA) ≥ 1,000 copies/mL.

Secondary endpoints are planned at W48 and W96.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age on the day of signing the informed consent.
* Be HIV-1 positive as determined according to national testing strategies
* Have a plasma HIV-1 RNA ≥1000 copies/mL within 30 days prior to the randomization,
* Have HIV treatment indication based on physician assessment according to local treatment guidelines
* Be naïve to antiretroviral therapy (ART) including investigational antiretroviral agents
* For women or transgender men of childbearing potential i.e. of childbearing age who are not menopausal, or permanently sterilized (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy) or not refraining from sexual activity: negative urinary test for pregnancy and acceptance to use contraceptive methods
* Understand the study procedures and voluntarily agree to participate by giving written informed consent for the trial.

Non-inclusion Criteria:

* Has ongoing (pulmonary or extra-pulmonary) tuberculosis
* Has any other history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.
* Is infected with HIV-2 or co-infected with HIV-1 and HIV-2
* Has received cabotegravir long acting or dapivirine pre-exposure prophylaxis (PrEP).
* Has received oral pre-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP) in the past three months or has had no negative HIV-1 serology performed
* Has documented or known resistance or possible resistance to study drugs (in France and where national guidelines recommend screening for primary resistance before starting first-line ART) as defined by the ANRS MIE AC43 Resistance group
* Has the following laboratory values at screening visit, within 30 days prior to the randomization:

  * AST (SGOT) and ALT (SGPT) >4.0 x upper limit of normal
  * Estimated glomerular filtration rate at time of screening <60 mL/min/1.73m², based on the CKD-EPI equation
* Has participated in a study with an investigational compound/device within 30 days prior to signing informed consent or anticipates participating in such a study involving an investigational compound/device during the course of this study.
* Has used systemic immunosuppressive therapy or immune modulators within 30 days prior to treatment in this study or is anticipated to need them during the course of the study
* Requires or is anticipated to require any of the prohibited or contraindicated medications noted in the trial protocol.
* Has significant hypersensitivity or other contraindication to any of the components of the study drugs.
* Is pregnant, breastfeeding, or expecting to conceive at any time during the study.
* Has any condition which might, in the investigator's opinion, compromise the safety of treatment and/or patient's adherence to study procedure.
* Is a person under guardianship or deprived of freedom by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of doravirine in combination with tenofovir and lamivudine as compared to dolutegravir in combination with tenofovir and lamivudine or emtricitabine in terms of virological efficacy at week 48 | Week 48
  The non-inferiority will be assessed in terms of virologic efficacy at week 48 under allocated treatment using the FDA snapshot algorithm (window period of 42-54 weeks), and measured by the proportion of subjects achieving a rate of HIV 1 RNA <50 copies/mL, in HIV-1 infected, treatment-naive subjects with pre-treatment viral load (HIV-1 RNA) ≥ 1,000 copies/mL.
  The rate of HIV 1 RNA will be measured by RT-PCR.

SECONDARY OUTCOMES:
Occurrence of obesity | Week 48; Week 96
  Obesity will be defined as having BMI≥30 kg/m² for Caucasian and African population and BMI≥27.5 kg/m² for Asian populations.
Occurrence of insulin resistance | Week 48; Week 96
  Proportion of subjects with newly measured HOMA≥2 as compared to baseline HOMA will be calculated with the following formula (glucose levels in mmol/L, insulin levels in mIU/L): HOMA =(glucose ×insulin)÷22.5
Occurrence of hypertension | Week 48; Week 96
  Proportion of subjects with hypertension newly detected compared to baseline. Hypertension will be defined as either being prescribed new anti-hypertension medication and/or by having diastolic blood pressure >90 mmHg AND/OR systolic blood pressure >140 mmHg during visit and confirmed during subsequent visit > 15 days after.
Non-inferiority of DOR in association with TDF and 3TC, compared to DTG in association with TDF and 3TC or FTC, in terms of virologic efficacy | Week 96
  Proportion of subjects in virologic success defined as achieving HIV-1 RNA <50 copies/mL at week 96 under allocated treatment using the FDA snapshot algorithm with a window period of 90 to 102 weeks; subjects not achieving viral success will be described according to the FDA snapshot recommendation
Occurrence of virological failures | Virological failure
  Proportion of confirmed virological failures. Virological failure will be defined as 1) confirmed HIV-1 RNA ≥ 200 copies/mL after initial response with HIV-1 RNA < 50 copies/mL at any time during the study or 2) non-response defined as either confirmed HIV-1 RNA ≥ 200 copies/mL at Week 24 or Week 36 (or any other unscheduled visit in-between) or confirmed HIV-1 RNA ≥ 50 copies/mL at Week 48, Week 72 and Week 96 (or any other unscheduled visit in-between).
Occurrence of HIV-1 drug resistances in patients with confirmed virological failure | Virological Failure
  Frequency of HIV-1 drug resistances in participants with a confirmed virological failure.
  Drug resistances will be defined according to the last version of the ANRS algorithm and to the last version of the Stanford algorithm.
Virological efficacy at a threshold of HIV 1 RNA<200 copies/mL | Week 48; Week 96
  Proportion of subjects achieving HIV 1 RNA<200 copies/mL under allocated treatment
Virological efficacy at a threshold of HIV 1 RNA<1000 copies/mL | Week 48; Week 96
  Proportion of subjects achieving HIV 1 RNA<1000 copies/mL under allocated treatment
Effect of baseline RT and integrase mutations on virological response | Week 48; Week 96
  Frequency of RT and integrase mutations at baseline and impact on the virological response
Occurrence of combined overweight and obesity | Week 48; Week 96
  Combined overweight and obesity will be defined as having BMI≥25 kg/m² for Caucasian and African populations and BMI≥23 kg/m² for Asian populations
Occurrence of weight gain ≥10% absolute body weight | Week 48; Week 96
  Proportion of subjects with ≥10% absolute weight gain from baseline
Changes in absolute weight gain | Week 48; Week 96
  Absolute weight gain will be calculated by simply subtracting the follow-up weight from baseline weight measured according to protocol procedures
Occurrence of diabetes | Week 48; Week 96
  Proportion of subjects with diabetes newly detected compared to baseline. Diabetes will be defined as either being prescribed new medication for diabetes mellitus and/or having a fasting glycemia ≥1.26 g/L during visit and confirmed during subsequent visit > 15 days after and/or in a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥ 200 mg/dL (11.1 mmol/L).
Safety and tolerability | Week 48; Week 96
  Any adverse event of any grade and those graded 3-4
Changes in waist circumference, hip circumference and waist-to-hip ratio | Week 48; Week 96
  Change from baseline in waist and hip circumferences and waist-to-hip ratio
Changes in fasting glycemia and insulin | Week 48; Week 96
  Change from baseline in fasting glycemia and insulin
Changes in fasting serum lipids | Week 48; Week 96
  Change from baseline in fasting serum lipids. The fasting serum lipids analyzed will be total cholesterol, HDL, LDL and triglycerides.
Changes in estimated glomerular filtration rate | Week 48; Week 96
  Change from baseline in estimated glomerular filtration rate. Estimated glomerular filtration rate (eGFR) will be calculated using the CKD-EPI equation
Occurrence of cardiovascular abnormalities | Week 48; Week 96
  Change from baseline in cardiovascular parameters (blood pressure profile, electrocardiographic and echocardiographic damages). These cardiovascular parameters assessments will be measured through an electrocardiogram, a transthoracic echocardiography and an ABPM, a 24-hour blood pressure Holter.
Changes in liver steatosis and clinically significant fibrosis | Week 48; Week 96
  Change from baseline in mean patient CAP and LSM measurements and occurrence of: Liver steatosis defined by CAP ≥ 263 dB/m2, and clinically significant liver fibrosis and cirrhosis defined by LSM ≥ 8.0 kPa and LSM ≥ 12.5 kPa, respectively
Occurrence of metabolic dysfunction-associated steatotic liver disease (MASLD) and metabolic-associated steatohepatitis (MASH) | Week 48; Week 96
  Change from baseline in mean patient CAP and LSM measurements and occurrence of: MASLD defined by the presence of liver steatosis with at least one cardiometabolic risk-factor (overweight/obesity; pre-or diabetes; hypertension; hypertriglyceridemia or low-HDL; and MASH defined by the presence of at least CSF in people with MASLD.
Changes in liver diseases biomarkers | Week 48; Week 96
  Changes from baseline in Fib-4, VCTE and FAST scores and presence at baseline or occurrence of: CSF defined as Fib-4 ≥ 2.67 and FAST score > 0.67 (high probability of MASH)
Changes in mental health and quality of life outcomes | Week 24; Week 48; Week 96
  Change from baseline in EQ-5D-3L, HIVTSQ, DASS-21, PSQI, WHOQOL HIV-BREF scores
Occurrence of Acquired Immune Deficiency Syndrome (AIDS), tuberculosis, Immune Reconstitution Inflammatory Syndrome (IRIS) or death | Week 48; Week 96
  Proportion of subjects with AIDS (defined as having CDC stage 3/C or WHO stage 4), tuberculosis, IRIS or death
Description of antiretroviral drugs trough plasma concentration in each arm | Week 4; Week 24; Week 48; Week 96
  DOR, DTG and M9 trough plasma concentration in samples taken pre-dose
Assessment of the effect of antiretroviral drugs trough plasma concentration on virological response | Week 4; Week 24; Week 48; Week 96
  DOR, DTG and M9 trough plasma concentration in samples taken pre-dose
Determining DOR, DTG and M9 trough plasma concentration thresholds predictive of virological response | Week 4; Week 24; Week 48; Week 96
  DOR, DTG and M9 trough plasma concentration in samples taken pre-dose
Assessment of the effect of antiretroviral drugs trough plasma concentration on safety endpoints | Week 4; Week 24; Week 48; Week 96
  DOR, DTG and M9 trough plasma concentration in samples taken pre-dose
Changes in CD4 cell count, CD4 percentage, CD8 cell count, CD8 percentage, CD4/CD8 ratio | Week 48; Week 96
  Change from baseline in CD4 cell count, CD4 percentage, CD8 cell count, CD8 percentage, CD4/CD8 ratio
Adherence to ART | Week 48; Week 96
  Adherence to ART by (1) pill count (considering a pill count adherence ratio <95% as sub-optimal adherence), (2) 4-days and 1-month recall questions at every trial visit, (3) by TFV-DP quantification in dried blood spots (LC/MS). ARV pill burden will also be an endpoint in order to study the relation between adherence and ARV pill burden.
Description of the distribution of CYP3A5/4 mutations according to ARV regimen | Study long
  Type and frequency of alleles variants in the gene coding for CYP3A5/4
Assessment of the impact of CYP3A5/4 mutations on PK | Study long
  Impact of CYP3A5/4 mutations on pharmacokinetics of DOR, DTG and M9
Assessment of the impact of CYP3A5/4 mutations on virological response and side effects | Study long
  Virological response and side-effects depending on CYP3A5/4 mutations
Explore additional polymorphism (i.e. UGT1A1) according to literature update | Baseline
  Assess additional polymorphism of UGT1A1
Cost-effectiveness and budget impact of using DOR-based versus DTG-based antiretroviral regimens | Study long
  Cost-effectiveness measured by (1) Incremental health benefits of using one regimen compared to the other (in DALYs and QALYs), (2) Incremental economic costs of using one regimen compared to the other (USD), (3) Budget impact of changing from one regimen to the other (USD)
Changes in truncal fat distribution in a sub-group of cisgender women enrolled in the trial | Week 48; Week 96
  Change from baseline in truncal fat distribution. Truncal fat repartition will be measured by the proportion of fat tissue using DEXA-scanner assessment
Changes in adipose tissue markers and immune activation markers in a sub-group of cisgender women enrolled in the trial | Week 48; Week 96
  Change from baseline in adipose tissue markers (adiponectin, leptin) and immune activation markers (sCD14, sCD163). Measurement will be made on stored serum samples by immunonephelometry or ELISA.
Changes in fat quality in a sub-group of cisgender women enrolled in the trial | Week 48
  Change from baseline (by abdominal subcutaneous surgical biopsy) in fat pathology, gene expression and global transcriptome analysis (RT-PCR and RNAseq). Measurement will be made on an abdominal fat tissue biopsy sample fixed for immunohistochemistry (Red Sirius, collagen 6, fibronectine, TFG-beta, alpha-SMA) and frozen for gene expression analysis by RT-PCR of markers of adipogenesis (PPARG, CEPBA), beiging (PRDM16, PGC1A), lipogenesis (FAS), adipocyte function (GLUT4), fibrosis (COL4, COL6, FN, TGFB, LOX, ASMA) and mDNA level (mDNA gene and nDNA).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SELLIER, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Beatriz GRINSZTEJN, Pr, Principal Investigator — INI-FIOCRUZ
Locations (19):
- Brazil (2):
  - Hospital Geral de Nova Iguaçu, Nova Iguaçu, Rio de Janeiro
  - Laboratory on Clinical research on AIDS-INI FIOCRUZ, Rio de Janeiro, Rio de Janeiro
- Hôpital Central de Yaoundé, Yaoundé, Cameroon
- Côte d’Ivoire (3):
  - Centre de prise en charge de Recherche et de Formation (CEPREF), Abidjan
  - Centre Médical de Suivi des Donneurs de Sang (CMSDS) - Centre National de Transfusion Sanguine (CNTS), Abidjan
  - CHU de Treichville, Service des Maladies Infectieuses et Tropicales (SMIT), Abidjan
- France (9):
  - CHU Bordeaux Pellegrin - Service des Maladies Infectieuses et Tropicales, Bordeaux
  - CHU Bordeaux St André - Service de Médecine Interne, Bordeaux
  - CHU Montpellier - Hôpital La Colombière - Service des Maladies Infectieuses et Tropicales, Montpellier
  - CHU Nantes Hôtel Dieu - Service des Maladies infectieuses et tropicales, Nantes
  - AP-HP Hôpital Lariboisière - Service de Maladies Infectieuses et Tropicales, Paris
  - AP-HP Hôpital Saint Louis - Service des Maladies Infectieuses et Tropicales, Paris
  - AP-HP Hôpital Saint Antoine - Service des Maladies Infectieuses et Tropicales, Paris
  - AP-HP Hôpital Pitié Salpêtrière - Service des Maladies Infectieuses et Tropicales, Paris
  - AP-HP Bichat Claude Bernard - Service des Maladies Infectieuses et Tropicales, Paris
- Centro de Saúde 1o de Maio, Maputo, Mozambique
- Thailand (3):
  - Chiangrai Prachanukroh, Chiang Rai
  - Lampang Hospital Internal Medicine department, Lampang
  - Phayao Hospital Internal Medicine department, Phayao

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] L'hostellier A, Kouanfack C, Chazallon C, Wagner-Cardoso S, Eholie SP, Banze N, Halue G, Capeau J, Delaugerre C, Moh R, Bonnet F, Mfeukeu Kuate L, Jaquet A, Perazzo H, Bernard C, Bastard JP, Goldwirt L, Vilquin P, Nhassengo PP, Lavalee M, Minvielle N, Dodd PJ, Marcy O, Molina JM, Grinsztejn B, Sellier PO. Doravirine versus dolutegravir-based regimen in antiretroviral treatment-naive people living with HIV-1 (ANRS0392s ELDORADO): protocol for an international, open-label, randomised, non-inferiority, phase III trial. BMJ Open. 2026 Feb 5;16(2):e110560. doi: 10.1136/bmjopen-2025-110560. PMID 41644158